CLINICAL TRIAL: NCT02952521
Title: Paired Biopsies to Develop a Cellular Signature
Brief Title: Ovarian Tumor Biopsies to Study Response to Treatments
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: KINOME
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Whole blood samples
  * Tumor tissue samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Epithelial ovarian cancer: * Whole blood sample collection
  * Up to 3 fresh tumor tissue core biopsies
  * Tumor tissue sample taken from tumor tissue already removed from surgery (if surgery is planned)
  Interventions: Procedure: Blood Draw; Procedure: Tumor Tissue Biopsy

INTERVENTIONS:
Procedure: Blood Draw — CA125 and ctDNA
Procedure: Tumor Tissue Biopsy — Only collected at time of surgery if patient undergoes surgical debulking

SUMMARY:
This is a research study to look at differences in tumor tissue from ovarian cancer patients that may help to determine response and resistance to treatments.

DETAILED DESCRIPTION:
Ovarian cancer participants will be asked to have two tumor biopsies during the research study. The first biopsy will be done prior to receiving the participants' assigned treatments as a part of their cancer care and the second biopsy will be done about 3-7 days after starting treatment. Participants who will undergo neoadjuvant treatment and then surgery, will also have their tumor tissue collected during surgery. Participants whose disease worsens while on treatment will also be asked to have an additional, optional tumor biopsy.

The tumor tissue samples will be studied to look at certain proteins and enzymes, including enzymes called kinomes, that may be important in determining response and resistance to the treatment that participants will receive as a part of their cancer care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Histological diagnosis of epithelial ovarian cancer
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Life expectancy of greater than 3 months
* Diagnosis of epithelial ovarian cancer undergoing chemotherapy as part of standard care or a clinical trial OR receiving a targeted therapy with a targeted agent
* Must be agreeable to paired biopsies
* Must have disease amenable to paired biopsy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Any contraindication to biopsy
* Need for anticoagulation that cannot be interrupted

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histological diagnosis of epithelial ovarian cancer
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Pearson correlation for changes between kinome and CA125 | 5 years
Paired T-test for differences in kinome between responders and non-responders | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No